CLINICAL TRIAL: NCT00351104
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Phase III Study of the Efficacy, Tolerability and Safety of Ketoprofen Topical Patch, 20% (KTP) in the Treatment of Pain Associated With Grade 1 or Grade 2 Ankle Sprain or Strain
Brief Title: Efficacy and Safety of Ketoprofen Topical Patch 20% in the Treatment of Pain Associated With Ankle Sprain or Strain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Stephen McMorn, Endo Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3269-301
Record Dates: First submitted 2006-06-30; First posted 2006-07-12 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Sprain; Strain
Keywords: Sprain; Strain; Pain; Ankle Pain; Muscle, Bone and Cartilage Disorders
MeSH Terms: conditions — Sprains and Strains; Pain; Cartilage Diseases

INTERVENTIONS:
Drug: Ketoprofen Topical Patch 20%

SUMMARY:
The purpose of this study is to evaluate the effect of a ketoprofen topical patch on the pain associated with ankle sprain or strain.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel group study will be conducted in patients with Grade 1 or Grade 2 ankle sprains or strains. Eligible patients will be randomized (in a 1:1 ratio) to receive double-blind treatment with either the KTP or a matching placebo patch to be applied once daily for 14 days. Patients will return to the clinic for assessments on Day 3, Day 7 and Day 14; a follow-up assessment will be conducted by telephone on Day 28. At each visit through Day 14, patients will rate their average pain intensity during daily activities and while at rest using an 11-point scale, and will rate their functional disability. Patients will also complete an electronic diary in which pain intensity and pain relief ratings will be recorded three times daily. Ratings of the quality of sleep will be recorded in the diary each morning, and the use of study treatment and rescue medication will be recorded in the diary each day. Ibuprofen will be provided as rescue medication

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* Diagnosis of Grade I or Grade II ankle sprain or strain
* Meet pain entry criteria
* Willing to discontinue use of any pain medication not provided as part of the study

Exclusion Criteria:

* Have a Grade 3 sprain or Grade 3 strain, bilateral sprain or strain, or concomitant fracture or wound at the site of the sprain or strain.
* Have received corticosteroids in the 30 days preceding screening
* Have a history or physical examination finding that is incompatible with safe participation in the study
* Have a history or physical examination finding that is incompatible with study product use
* Are taking medications or other substances contraindicated due to the nature of the study medication or the potential for drug interactions.
* Are taking medications that may significantly affect renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Average pain intensity during daily activities

SECONDARY OUTCOMES:
Average pain intensity while at rest; Functional disability; Use of rescue medication; Quality of sleep; Patient's and physician's global assessments of study medication

CONTACTS AND LOCATIONS:
Overall Officials: PPD, Principal Investigator — PPD Austin, TX
Locations (1):
- PPD, Austin, Texas, United States